CLINICAL TRIAL: NCT02425605
Title: Efficacy of Localized Concurrent Chemo-radiation Therapy and Sorafenib Sequential Therapy in Advanced Hepatocellular Carcinoma: a Prospective Phase 2 Trial
Brief Title: Efficacy of Localized Concurrent Chemo-radiation Therapy and Sorafenib Sequential Therapy in Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0803
Record Dates: First submitted 2015-04-14; First posted 2015-04-24 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CCRT-sorafenib group (Experimental)
  Interventions: Radiation: CCRT; Drug: sorafenib

INTERVENTIONS:
Radiation: CCRT — The subject is treated with a total of 45 Gy of external beam radiotherapy (1.8 Gy per session, 5 sessions a week, for 5 weeks), with hepatic arterial infusion of 5-flourouracil (5-FU) during the first and last 5 days of radiation therapy (5-FU 500 mg infusion for 5 hours) for radiosensitization through the pre-inserted chemoport.
  Other Names: Localized concurrent chemoradiation therapy(CCRT)
Drug: sorafenib — Four weeks after completion of CCRT, the subject is given daily sorafenib treatment and will be followed for survival.
  Other Names: sorafenib(Nexavar®) sequential therapy

SUMMARY:
This is a single-center, single-arm, open-label, prospective phase 2 trial to assess the efficacy of localized concurrent chemoradiation therapy (CCRT) and sorafenib sequential therapy in subjects with advanced HCC. Approximately 47 subjects will be enrolled and will receive CCRT and sorafenib sequentially until all-cause mortality.

DETAILED DESCRIPTION:
This is a single-center, single-arm, open-label, prospective phase 2 trial to assess the efficacy of localized concurrent chemoradiation therapy (CCRT) and sorafenib sequential therapy in subjects with advanced HCC. Approximately 47 subjects will be enrolled and will receive CCRT and sorafenib sequentially until all-cause mortality.

Sorafenib is the current standard of care for advanced hepatocellular carcinoma (HCC) patients following clinical results from the two pivotal trials in Western and Asian patients. The median overall survival in patients with unresectable hepatocellular carcinoma (HCC) who are treated with sorafenib have shown to be approximately 14 months. However in the presence of portal vein invasion or extrahepatic metastases, the median overall survival is significantly lowered to 5.6 - 8.9 months.

Going forward, improvement in patient-related outcomes would be highly desirable.

A pilot study has been conducted in subjects with advanced HCC with portal vein invasion for which effective therapeutic methods have not been established. This was a single-center, open-label study of localized concurrent chemoradiation therapy (CCRT) for locally advanced HCC patients with portal vein invasion. A total of 40 subjects with advanced HCC with portal vein invasion were enrolled. The subjects were treated with a total of 45 Gy of external beam radiotherapy (1.8 Gy per session, 5 sessions a week, for 5 weeks), with hepatic arterial infusion of 5-flourouracil (5-FU) during the first and last 5 days of radiation therapy (5-FU 500 mg infusion for 5 hours) through the pre-inserted chemoport. Eighteen (45%) subjects had an objective tumor response at 1 month after completion of localized CCRT. The 3-year survival rate was 24.2% and median overall survival was 13.1 months.

Treatment-related serious adverse events (CTCAE grade 3 or higher) were anemia, leukopenia, thrombocytopenia, mucositis and liver decompensation, and their rates were 2.5%, 2.4-5.0%, 17.5%, 10% and 7.3-17.5%, respectively. In addition, 2.4-5.0% of adverse events were chemoport-related adverse events including infection and port obstruction.

Although sorafenib has been shown to increase overall survival in advanced HCC patients as compared to placebo through anti-angiogenesis effect, its tumoricidal effect is not evident. Meanwhile, based on the above analysis from the pilot study, localized CCRT has been regarded as a promising treatment with tumoricidal effect for advanced HCC patients. Therefore, combining sorafenib treatment with CCRT is anticipated to augment anti-tumor effect and improve tumor response and median overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have confirmed diagnosis of unresectable hepatocellular carcinoma (HCC) categorized to stage C based on Barcelona Clinic Liver Cancer (BCLC) staging system with any of following criteria: 1) Lesion limited to a single lobe that is within the radiotherapy field, 2) Lesion not limited to a single lobe, but the lesion that is not within the radiotherapy field can be controlled by transarterial chemoembolization or radiofrequency ablation, 3) Presence of metastatic lesions that measure < 1.0 cm in the long axis, 4) The lesion can be accurately measured in at least one dimension as ≥ 1.0 cm
* Males or females aged at least 20 years and below 76 years
* Eastern Cooperative Oncology Group performance status (ECOG-PS) 0 or 1
* Adequate liver function, defined as: 1) Child-Pugh score ≤ 7, 2) Bilirubin ≤ 3.0 mg/dL
* Adequate bone marrow function, defined as: 1) Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, 2) White blood cell count (WBC) ≥ 4.0 × 109/L, 3) Platelet count ≥ 60 × 109/L
* Adequate renal function, defined as serum creatinine < 2.0 mg/dL
* Subjects with hepatitis B virus (HBV)-related HCC must have adequately controlled HBV replication status
* Adequate blood coagulation factors, defined as international normalized ratio (INR) ≤ 2.3
* Provide written informed consent
* Willing and able to comply with all aspects of the protocol

Exclusion Criteria:

* Significant liver function impairment, defined as bilirubin > 3.0 mg/dL or uncontrolled ascites
* Imaging findings for HCC corresponding to any of the following: 1) Diffuse HCC with > 50% liver occupation, that is not adequate for external radiotherapy, 2) Presence of metastatic lesions that measure ≥ 1.0 cm in the long axis
* Uncontrolled significant active infection
* Presence of active malignancy (except for HCC)
* Females who are lactating or pregnant; females of childbearing potential who have not received pregnancy test or shown positive on pregnancy test
* Any medical or other condition that in the opinion of the investigator would preclude the subject's participation in a clinical study
* Major surgery within 4 weeks prior to enrollment

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-12-03; Primary Completion 2017-09-22 (Actual); Study Completion 2017-09-22 (Actual)

PRIMARY OUTCOMES:
Overall survival | 36 months after the enrollment

SECONDARY OUTCOMES:
PFSL defined as dynamic CT scan | 36 months after the enrollment
  Progression-free survival in the liver(PFSL)
PFSO defined as definitive imaging technique | 36 months after the enrollment
  progression-free survival overall (PFSO)
tumor response defined as modified RECIST | 36 months after the enrollment
toxicity defined as NCI-CTC(version 4.02) | 36 months after the enrollment
  toxicity defined as National Cancer Institute-Common Toxicity Criteria (version 4.02)

CONTACTS AND LOCATIONS:
Overall Officials: Beom Kyung Kim, M.D., Ph.D., Principal Investigator — Severance Hospital
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea